CLINICAL TRIAL: NCT07063238
Title: A Double-Blind, Placebo-Controlled and Active-controlled Trial to Evaluate the Effect of a Supratherapeutic Dose of MK-8527 on the QTc Interval in Healthy Adult Participants
Brief Title: A Clinical Study of MK-8527 in Healthy Adult Participants (MK-8527-014)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 8527-014; MK-8527-014 (Other: MSD)
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Healthy
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MK-8527 PLUS Moxifloxacin and Placebo (Experimental): Participants receive a single dose of MK-8527 followed by a single dose of moxifloxacin and a single dose of placebo depending on randomization.
  Interventions: Drug: MK-8527; Drug: Moxifloxacin; Drug: Placebo
- Moxifloxacin PLUS MK-8527 and Placebo (Experimental): Participants receive a single dose of moxifloxacin followed by a single dose of MK-8527 and a single dose of placebo depending on randomization.
  Interventions: Drug: MK-8527; Drug: Moxifloxacin; Drug: Placebo
- Placebo PLUS MK-8527 and Moxifloxacin (Experimental): Participants receive a single dose of placebo followed by a single dose of MK-8527 and a single dose of moxifloxacin depending on randomization.
  Interventions: Drug: MK-8527; Drug: Moxifloxacin; Drug: Placebo

INTERVENTIONS:
Drug: MK-8527 — Oral administration
Drug: Moxifloxacin — Oral administration
Drug: Placebo — Oral administration

SUMMARY:
Researchers are looking for new medicines to prevent Human Immunodeficiency Virus Type 1 (HIV-1) infection. HIV-1 is the most common type of HIV, which is a virus that attacks cells of the immune system. Medicines to prevent HIV-1 infection are called pre-exposure prophylaxis (PrEP). Some people may have trouble following a PrEP plan because it involves either taking medicine everyday by mouth or getting injections (shots) often.

MK-8527 is a study medicine designed to prevent HIV-1 infection. MK-8527 is different from standard (usual) PrEP because it is taken once a month, by mouth, as a tablet.

The goal of this study is to learn if taking a higher-than-normal dose of MK-8527 increases the QT interval (a measure of heart rhythm) by a certain amount.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Is in good health before randomization
* Has body mass index (BMI) between 18 and 32 kg/m^2, inclusive

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has history of clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological abnormalities or diseases.
* Has history of cancer (malignancy).
* Has positive test(s) for Hepatitis B surface antigen (HBsAg), hepatitis C antibodies or human immunodeficiency virus (HIV).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2025-08-12 (Actual); Primary Completion 2025-12-06 (Actual); Study Completion 2025-12-29 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in QT interval corrected for heart rate (QTc) following MK-8527 administration | Baseline and up to approximately 24 hours
  Change from Baseline in QTc following MK-8527 administration will be reported.

SECONDARY OUTCOMES:
Number of participants who experience one or more adverse events (AEs) | Up to approximately 7 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants that experience AEs will be reported.
Number of participants who discontinue study intervention due to an AE | Up to approximately 7 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants that discontinue study intervention due to an AE will be reported.
Change from Baseline in QTc following moxifloxacin administration | Baseline and up to approximately 24 hours
  Change from Baseline in QTc following moxifloxacin administration will be reported.
Area Under the Plasma Concentration-Time curve From Time 0 to 24 hours (AUC0-24) of MK-8527 | At designated timepoints (up to 24 hours postdose)
  Blood samples will be collected at multiple time points to estimate AUC0-24 of MK-8527
Area Under the Plasma Concentration-Time curve From Time 0 to 168 hours (AUC0-168) of MK-8527 | At designated timepoints (up to 168 hours postdose)
  Blood samples will be collected at multiple time points to estimate AUC0-168 of MK-8527
Area Under the Plasma Concentration-Time curve From Time 0 to infinity (AUC0-inf) of MK-8527 | At designated timepoints (up to approximately 7 weeks)
  Blood samples will be collected at multiple time points to estimate AUC0-inf of MK-8527
Maximum plasma concentration (Cmax) of MK-8527 | At designated timepoints (up to approximately 7 weeks)
  Blood samples will be collected at multiple time points to estimate Cmax of MK-8527
Time to maximum plasma concentration (Tmax) of MK-8527 | At designated timepoints (up to approximately 7 weeks)
  Blood samples will be collected at multiple time points to estimate Tmax of MK-8527

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Hassman Research Institute Marlton Site ( Site 0001), Marlton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com